CLINICAL TRIAL: NCT00592215
Title: A Pilot Study of Mifepristone Followed by Misoprostol in Women Undergoing Second Trimester Abortion
Brief Title: Second Trimester Labor Induction
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00010268; 2007-663
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Second Trimester Labor Induction
Keywords: Second trimester labor induction
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Mifepristone followed by labor induction with misoprostol after 6-8 hours
  Interventions: Drug: Experimental (mifepristone and misoprostol)

INTERVENTIONS:
Drug: Experimental (mifepristone and misoprostol) — Mifepristone 200mg followed by labor induction with misoprostol after 6-8 hours

SUMMARY:
A superior second trimester medical abortion regimen has not been identified. Studies suggest that a regimen of mifepristone and misoprostol given 36 to 48 hours apart has the shortest median induction-to-abortion interval, highest 24-hour abortion rate, and low rates of adverse events. Narrowing the interval between the two medications without clinically reducing effectiveness may increase access and acceptability for patients and reduce costs. Data from studies on first trimester abortions suggest that the 6 to 8 hour interval between mifepristone and misoprostol is as efficacious as the 36 to 48 hour interval. There are no studies on shorter intervals with same day administration between mifepristone and misoprostol in second trimester abortions.

The primary objective is to assess the efficacy of the combined mifepristone/misoprostol regimen for abortions between 17 0/7 and 23 6/7 weeks' gestation using an interval of 6 to 8 hours between the two medications.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking women
* 18 years of age and above
* Voluntarily choose to undergo pregnancy termination via labor induction
* An ultrasound-confirmed singleton intrauterine pregnancy between 17 0/7 and 23 6/7 weeks gestation
* Able to provide written consent

Exclusion Criteria:

* Premature rupture of membranes
* Preterm labor
* Intrauterine fetal demise
* Chronic systemic corticosteroid use or adrenal disease
* Hypersensitivity to prostaglandins
* Cardiovascular disease such as angina, valvular disease, arrhythmia, cardiac failure
* Known coagulopathy or treatment with anticoagulants
* Prior caesarean delivery or myomectomy
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Abortion rate | 8 hours after misoprostol administration

CONTACTS AND LOCATIONS:
Overall Officials: Rameet Singh, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland